CLINICAL TRIAL: NCT04743921
Title: Eﬀects of Reparel™ Knee Sleeve on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amit Momaya, Assistant Professor, Section Chief, Sports Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300006549
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Reparel Sleeve Group (Experimental): Patients receiving reparel knee sleeve for treatment of knee osteoarthritis.
  Interventions: Device: Reparel Knee Sleeve

INTERVENTIONS:
Device: Reparel Knee Sleeve — Patients who are recommended for non-operative management of knee osteoarthritis and have been consented in clinic to participate in the study will be given a Reparel™ knee sleeve to wear for knee osteoarthritis management. Each device will be numbered and recorded in the patient's REDCap entry for future reference if needed. Following administration of the Reparel™ knee sleeve, patients will be given instructions on how to use/wear the sleeve while performing activities of daily living or sports that had previously resulted in knee pain and also be asked to do the follows: wear the sleeve as much as they possibly can; not change their usual activities and diet during the time they are on this study; record in a diary the number of hours sleeve was worn per day; record any adverse eﬀects or discomfort due to sleeve use; refrain from altering treatment for knee osteoarthritis.

SUMMARY:
The goals of treating knee osteoarthritis (OA) is to improve or maintain quality of life, mobility and function, pain relief, and improve inﬂammation. The diﬀerent treatment options for knee OA have been extensively studied and implemented, but the optimum treatment is still undecided. There is a belief that anti-inﬂammatory sleeve technology may be beneﬁcial in treating knee OA. The purpose of this study is to determine the clinical eﬀects of Reparel™ knee sleeve regarding mobility, functionality, and pain outcomes in managing knee OA.

DETAILED DESCRIPTION:
Standard knee compression sleeves have been described throughout literature to provide beneﬁts in pain and functional outcomes through support of the ligamentous structures. Bracing is both an eﬀective and economical treatment for osteoarthritis and serves as a crucial option in the treatment of knee OA to aid in both delaying surgery and as options for young patients, or patients that are not ideal surgical candidates. Although knee sleeves are commonly utilized treatment modalities, there is a signiﬁcant paucity of literature on the eﬀects of thermo-active braces in the treatment of knee OA. This investigation will examine this non-operative treatment modality and study it eﬀect for the treatment of knee OA specifically by investigating the Reparel Knee Sleeve. The Reparel Knee Sleeve is a Class I Medical Device (510(k) exempt) and used in general sports medicine practice for the alleviation of knee pain. The authors expect that the Reparel thermos-active knee sleeve will have a signiﬁcant eﬀect on pain relief from knee OA.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis visible on knee radiograph
* patient opting for non-surgical treatment
* no corticosteroid knee injection for 90 days prior to consent
* no corticosteroid knee injection for 90 days following consent

Exclusion Criteria:

* bilateral symptomatic knee osteoarthritis
* prior surgery on the knee of interest
* hardware present on the knee of interest
* gross instability detected on physical exam
* malignancy in the knee of question

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Momaya, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reparel Sleeve Group
Started | 14
Completed | 13
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Average age and standard deviation was calculated for males and females separately
  years
    Female: number analyzed (Participants) | 10
    Female | 60.5 (12.8)
    Male: number analyzed (Participants) | 4
    Male | 66.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter squared] — Population: There were a total of 14 participants: 4 males and 10 females.
  kilograms per meter squared
    Male: number analyzed (Participants) | 4
    Male | 33.7 (2.6)
    Female: number analyzed (Participants) | 10
    Female | 34.3 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: University of California, Los Angeles (UCLA) Activity Score
Description: This is a questionnaire that measures current activity level. Patients self report their current activity level. It ranges from 1-10. A patient scoring themselves as a 1 is the lowest current activity level and represents someone who is wholly inactive. A patient scoring themselves as a 10 is the highest current activity level and represents someone able to regularly participate in impact sports.
Time Frame: 3 months
Population: Although 14 patients were enrolled at baseline, only 12 patients filled out their surveys at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 5.4 (1.4)

2. Primary Outcome: Lysholm Score
Description: This is a questionnaire that is self-reported by the patient. It is meant to measure a patient's ability to manage activities of daily living as it relates to their knee. The score range is from 0 to 100. A score of 0 is the lowest score associated with lower ability to manage activities of daily living, and a score of 100 is the highest score associated with a higher ability to manage activities of daily living.
Time Frame: 3 months
Population: Although 14 patients were enrolled at baseline, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 75.0 (15.3)

3. Primary Outcome: Oxford Knee Score (OKS)
Description: This is a questionnaire that is self-reported by the patient. It measures knee pain and function. It is scored from 0 to 48. A score of 0 represents the lowest score and is associated with higher knee pain and lower function. A score of 48 represents lower knee pain and higher function.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 38.2 (7.0)

4. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score Pain (KOOS-P)
Description: This is a patient questionnaire that is self-reported. It is a measure of how much pain a patient has during different activities. A score of 100 represents the lowest level of pain with different activities. A score of 0 represents the highest amount of pain with different activities.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 72.9 (15.2)

5. Primary Outcome: Single Assessment Numeric Evaluation (SANE)
Description: This is a patient questionnaire that is self-reported by the patient. It represents a patient's perceived functional level of their affected joint as a percentage of normal. The score is ranged from 0% to 100%. A score of 100% is the best outcome with the patient perceiving their functional level as 100% of normal.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: percentage score
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
percentage score | 72.0 (31.0)

6. Primary Outcome: Visual Analog Scale (VAS)
Description: This is a patient questionnaire that is self-reported by the patient. It measures how much knee pain the patient is having. The score ranges from 0 to 10. A score of 0 represents the best outcome with the least amount of pain. A score of 10 is the worst outcome with the most amount of pain.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 3.0 (2.9)

7. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score Symptoms (KOOS-Sy)
Description: This is a patient questionnaire that is self-reported. It represents the amount of knee symptoms a patient has. A score of 0 represents the worst outcome with a patient reporting the most symptoms. A score of 100 represents the best outcome with patients reporting the least symptoms.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 75.6 (16.1)

8. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score Activities of Daily Living (KOOS-ADL)
Description: This is a patient questionnaire that is self-reported by the patient. It measures the ability of a patient to perform activities of daily living as it relates to a patient's knee. A score of 0 represents the worst outcome with patients reporting the most difficulty performing activities of daily living. A score of 100 represents the best outcome with patients reporting the least difficulty with performing activities of daily living.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 patients filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 81.37 (16.0)

9. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score Quality of Life (KOOS-QOL)
Description: This is a patient questionnaire that is self-reported by the patient. It measures a patient's quality of life as it relates to their knee. A score of 0 represents the lowest quality of life as it relates to a patient's knee. A score of 100 represents the highest quality of life as it relates to a patient's knee.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 59.9 (21.6)

10. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score Sports and Recreation (KOOS-Sp)
Description: This is a patient questionnaire that is self-reported by the patient. It measures a patient's ability to perform sports and recreation as it relates to their knee. A score of 0 represents the lowest ability to perform sports and recreation as it relates to their knee. A score of 100 represents the highest ability to perform sports and recreation as it relates to their knee.
Time Frame: 3 months
Population: Although 14 patients were enrolled, only 12 filled out their questionnaires at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparel Sleeve Group
Number analyzed (Participants) | 12
score on a scale | 47.5 (21.3)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Reparel Sleeve Group
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 6/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reparel Sleeve Group (N=14)
Knee swelling (Skin and subcutaneous tissue disorders) | 3 — 3 patients experienced knee swelling after 2 weeks
Skin Irritation (Skin and subcutaneous tissue disorders) | 2
Lower leg and foot swelling (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT04743921/Prot_SAP_001.pdf